CLINICAL TRIAL: NCT07239557
Title: Optimal Interval for Periodic Alveolar Recruitment Maneuvers Achieving 90% Lung Re-expansion During Intraoperative Mechanical Ventilation: A Randomized Biased-Coin Sequential Trial
Brief Title: Optimal Interval for Periodic Alveolar Recruitment Maneuvers Achieving 90% Lung Re-expansion During Intraoperative Ventilation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: E2025034
Record Dates: First submitted 2025-09-25; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Major Abdominal Surgery; Atelectasis; Lung-protective Ventilation; Lung Ultrasound Score; Postoperative Pulmonary Complications
Keywords: Laparoscopy; Trendelenburg position; Major abdominal surgery; Mechanical ventilation; Periodic recruitment maneuvers; Lung recruitment strategy; Respiratory function; Lung-protective ventilation; Lung ultrasound score; Effective concentration for 90% (EC90)
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PARM (Experimental)
  Interventions: Procedure: Different interval of PARM

INTERVENTIONS:
Procedure: Different interval of PARM — The initial time interval of PARM was 0.5 hours/time, and the different interval of PARM was assigned by random partial coin sequential method.If the previous patient did not respond to postoperative assessment of lung opening, the interval between expansion of the lungs was shortened by 10 minutes for the next patient; If lung opening is effective, there is an 11% chance that the next patient will have an 10-minute expansion interval and an 89% chance that the time interval will remain unchanged.

SUMMARY:
This study aims to determine the optimal interval for periodic alveolar recruitment maneuvers (PARM) that can achieve effective lung re-expansion in 90% of patients undergoing intraoperative mechanical ventilation during abdominal laparoscopic surgery in the low Trendelenburg position. Identifying the most effective frequency of PARM is crucial for establishing lung-protective ventilation strategies, with the ultimate goal of reducing intraoperative atelectasis, decreasing postoperative pulmonary complications, and accelerating recovery.

Patients are randomized using a biased-coin sequential design. PARM is initially applied every 0.5 hours, and the effectiveness of lung re-expansion is evaluated before the end of surgery. The primary outcome is the effectiveness of recruitment, assessed by a combination of lung ultrasound scores and shunt fraction. Secondary outcomes include mechanical power at the end of surgery, time-weighted average mechanical power during ventilation, postoperative P/F ratio, dead space fraction, air test results, intraoperative adverse events, incidence of respiratory failure in the PACU and postoperative period, and postoperative length of stay.

This trial is expected to provide robust evidence for defining the optimal RM interval in protective ventilation protocols for patients undergoing laparoscopic abdominal surgery, thereby contributing to improved perioperative respiratory outcomes.

DETAILED DESCRIPTION:
This study is designed to evaluate the optimal interval of periodic alveolar recruitment maneuvers (PARM) to achieve effective lung re-expansion (defined as LUS ≤1 and shunt fraction <10%) in 90% of elderly patients undergoing laparoscopic anterior resection in low Trendelenburg position. This is a single-arm, biased-coin sequential design study. The initial PARM interval is 30 min, adjusted in 10 min increments based on response. The primary outcome is recruitment efficacy. Secondary outcomes include intraoperative mechanical power, P/F ratio, postoperative pulmonary complications, and length of hospital stay. This study aims to inform optimal RM intervals in protective ventilation protocols.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-80 years
* Undergoing elective laparoscopic anterior resection (expected mechanical ventilation duration 2-5 hours)
* Intermediate risk for postoperative pulmonary complications
* Room air SpO₂ ≥94%

Exclusion Criteria:

* History of pneumonia within 1 month or mechanical ventilation ≥1 hour
* Preoperative 12-zone LUS with any single zone score ≥2
* Preoperative shunt fraction ≥10%
* Progressive neuromuscular disease
* Severe emphysema/COPD or subpleural bullae ≥2 cm
* Intracranial hypertension
* Participation in other studies or refusal to participate

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of recruitment | Intraoperative
  The effectiveness of recruitment assessed by a combination of lung ultrasound scores and shunt fraction。At the end of surgery (with the patient in the supine position, after at least 5 minutes of apnea under mechanical ventilation without spontaneous breathing, and at the specified interval since the last recruitment maneuver), a lung ultrasound examination was performed. Lung re-expansion was considered effective if the 12-zone lung ultrasound score (LUS) was ≤1 per zone and the shunt fraction was <10%.

SECONDARY OUTCOMES:
Mechanical power at the end of surgery | With the patient in the supine position, after at least 5 minutes of apnea under mechanical ventilation without spontaneous breathing, and at the specified interval since the last recruitment maneuver
  Mean or median mechanical power
Time-weighted average mechanical power during surgery | During intraoperative mechanical ventilation
  Mechanical power per ventilation time
The P/F ratio at the end of surgery, | At the end of surgery (with the patient in the supine position, after at least 5 minutes of apnea under mechanical ventilation without spontaneous breathing, and at the specified interval since the last recruitment maneuver)
  P/F ratio = PaO₂ / FiO₂.Statistical measure: Incidence of P/F ratio ≤400. The P/F ratio is an objective research parameter, and a P/F ratio ≤400 indicates the presence of atelectasis.
Dead space rate | At the end of surgery (with the patient in the supine position, after at least 5 minutes of apnea under mechanical ventilation without spontaneous breathing, and at the specified interval since the last recruitment maneuver)
  Arterial carbon dioxide partial pressure (PaCO2); partial pressure of carbon dioxide in end expiratory gas (PetCO2); Dead space fraction = (PaCO2-PetCO2)/ PaCO2.
Air-breathing test | At the end of surgery (with the patient in the supine position, after at least 5 minutes of apnea under mechanical ventilation without spontaneous breathing, and at the specified interval since the last recruitment maneuver)
  After completion of ultrasound and arterial blood gas measurements, the inspired oxygen concentration was adjusted to 21%. SpO₂ was observed and recorded after 5 minutes.The incidence of a positive air-breathing test, defined as SpO₂ ≤96%, was recorded
Intraoperative hypotension | During mechanical ventilation in the intraoperative period.
  Defined as mean arterial pressure (MAP) <60 mmHg from any cause, lasting for more than 3 minutes。
Intraoperative vasopressor use. | During intraoperative mechanical ventilation
  Defined as any episode of MAP <60 mmHg during mechanical ventilation requiring the administration of catecholamine vasopressors, including dopamine, epinephrine, or norepinephrine. Occurrence of such an event was recorded as positive.
Intraoperative mild hypoxemia | During intraoperative mechanical ventilation
  SpO₂ ≤96% lasting for more than 3 minutes
Intraoperative severe hypoxemia | During intraoperative mechanical ventilation
  SpO₂ ≤92% lasting for more than 3 minutes
Lung ultrasound score (LUS) in the post-anesthesia care unit (PACU) | Awake with spontaneous breathing before discharge from the PACU
  The 12-zone lung ultrasound score (LUS) ranges from 0 to 3 per zone (total 0-36). Higher scores indicate more severe atelectasis.
Rate of respiratory failure at post-anesthesia care unit (PACU) | Stay in the PACU for at least 20 minutes and at most 3 hours; assessed at 5 to 10 minutes before leaving PACU
  PaO₂/FiO₂ <300 mmHg, or PaO₂ <60 mmHg or SpO₂ <90% while awake and breathing room air.
Rate of postoperative respiratory failure | Day1 to 5 after surgery
  PaO₂/FiO₂ <300 mmHg, or PaO₂ <60 mmHg or SpO₂ <90% while awake and breathing room air.
Rate of sustained hypoxaemia | Day 1 to 5 after surgery
  Sustained hypoxaemia, hypoxaemia at any two consecutive days; hypoxaemia: during a follow-up visit when the patient was awake and breathing room air, SpO2 ≤ 92% or the change of SpO2 (ΔSpO2, preoperative SpO2 minus postoperative SpO2) ≥ 5%.
Postoperative pulmonary complications, Grades 1-4 | Day 0 to 5 after surgery
  Operational Definitions of Postoperative Pulmonary Complications (Doi: 10.1001/jama.296.15.1851), graded on a scale from 1 to 4.
Postoperative pulmonary complications, Grades 2-4 | Day 0 to 5 after surgery
  Operational Definitions of Postoperative Pulmonary Complications (Doi: 10.1001/jama.296.15.1851), graded on a scale from 2 to 4
Pneumothorax | Day 0 to 7 after surgery
  Defined as the presence of air within the pleural cavity, with the visceral pleura not being surrounded by a vascular pattern.
Postoperative hospitalization days | Day 0 to 30 after surgery
  The duration between the operation date and the actual discharge date.
Unexpected admission to ICU | within 30 days after surgery
  It does not include the patients who enter ICU at the request of surgeons but have normal spontaneous breathing, stable circulation and no disturbance of consciousness.
Death from any cause | Day 0 to 30 after surgery
  Intraoperative or postoperative death from any cause

IPD SHARING:
Plan to Share IPD: No